CLINICAL TRIAL: NCT02878044
Title: Shared Decision Making in Patients With Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juan P. Brito Campana, MBBS, Assistant Professor of Medicine, Senior Associate Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-003809
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Thyroid Nodule; Thyroid Cancer
Keywords: Shared Decision Making, Decision Aid
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Arm (Experimental)
  Interventions: Other: Thyroid Decision Aid

INTERVENTIONS:
Other: Thyroid Decision Aid — The Thyroid Decision Aid is a tool designed to help clinicians and patients discuss treatment options for thyroid nodules.

SUMMARY:
The objective of this project is to evaluate a treatment decision aid for patients with low risk thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of low risk thyroid cancer

Exclusion Criteria:

-Does not have the cognitive capacity to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Distribution of treatment choices between patients receiving usual care versus decision aid | Up to six months
  Distribution of treatment choices between patients receiving usual care versus decision aid

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Brito Campana, MBBS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials